CLINICAL TRIAL: NCT05836298
Title: Impact of C-reactive Protein on Non Surgical Periodontal Treatment Performed With Mini-invasive Approach
Brief Title: Impact of C-reactive Protein on Non Surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 149-22-PO
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Each selected patient underwent randomly, without anaesthesia, after recording periodontal parameters, the two following treatments: in one, maxillary quadrants were treated as conventional Quadrant Scaling and Root Planing (SRP) or MINST treatment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis quadrant Scaling root planing (SRP) (Placebo Comparator): Each selected subject underwent quadrant SRP
  Interventions: Other: Non-surgical periodontal treatment
- MINST treatment (Active Comparator): Non surgical periodontal treatment performed with Minimally invasive non-surgical therapy (MINST) approach
  Interventions: Other: Non-surgical periodontal treatment

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Each selected patient underwent randomly, without anaesthesia, after recording periodontal parameters, the two following treatments: in one, maxillary quadrants were treated as conventional Quadrant Scaling and Root Planing (SRP) or MINST

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence the management of Periodontitis, the aim of this study was to evaluates, at 12-months follow-up, the post-treatment clinical and serum parameters in patients with periodontitis, treated by either Quadrant- Scaling and Root Planing (Q-SRP) treatment versus conventional Minimally invasive non-surgical therapy (MINST) treatment on serum C-reactive protein (CRP) and on Lipoprotein-associated phospholipase A2. Patients were also recalled for supportive periodontal treatment. The main objective was to analyze the effects of MINST or Q-SRP on clinical parameters and serum CRP and Lipoprotein-associated phospholipase A2 changes and if high CRP parameters at baseline influenced non surgical periodontal treatment.

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2016. The local ethical committee approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent. Subjects with a diagnosis of periodontitis were enrolled in this clinical trial. The inclusion criteria were: 1) good condition of general health, 2) a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm, 3) no involvement of the furcation, 4) a minimum of six teeth per quadrant, respectively. The exclusion criteria were: 1) periodontal therapy during the last 12 months, 2) assumption of antibiotics during the last 6 months, 3) pregnancy, 4) any systemic condition which might affect the effects of the study treatment, 5) previous or current radiation or immunosuppressive therapies, 5) use of mouthwash containing antimicrobials during the previous 3 months, 6) no use of hormonal contraceptives, 7) medication by anti-inflammatory and immunosuppressive drugs, 8) previous history of hard-drinking, 9) smoking, 10) class II and III tooth mobility. The primary outcome was the analysis of NSPT performed with either MINST or Q-SRP on periodontal parameters and tooth loss and on serum CRP expression changes between groups after 1- and also 8 years. Furthermore, The secondary objective was to examine the influence and interaction between NSPT protocol (MINST used as a reference) and the duration of treatment on serum CRP changes, as well as whether high baseline CRP levels influenced the efficacy of NSPT after 1-year follow-up. Variations for PD, CAL, FMBS, FMPS, PISA, Lp-PLA2 and CRP were collected and analyzed at 1, 3-, 6-month and at 1-year follow-up.

Patients randomly undergo Q-SRP or MINST non surgical periodontal treatment performed in one session.

All patients underwent an initial session with supragingival debridement. In addition, they received detailed information about the aetiology of periodontitis and individualized oral hygiene instructions, which included inter-dental plaque control and toothbrushing using a modified Bass technique. All participants were provided with the same type of toothbrush and toothpaste§ as well as interdental brushes‖.

The NSPT was achieved by both hand and ultrasonic instrumentation using a No. 5/6/7 tip according to operator preference. In both groups, the ultrasonic device was used with constant water irrigation and with a 20 Hz of frequency at a 60 µn power setting. Patients in the Q-SRP group received quadrant scaling in four different sessions with an interval of 1 week between each quadrant treatment session. Each patient's first session started in the upper right maxillary quadrant.

MINST was performed under local anaesthesia through careful subgingival debridement using ultrasonic scalers with specific thin tips# and Gracey micro-curettes** to minimize the trauma for the soft tissues. Under 3.5x magnification loupes, supra- and subgingival deposits were thoroughly debrided. After the operation, there was no subgingival rinsing to promote the establishment of a stable blood clot.

No mouthwashes, antibiotics or other drugs were prescribed after treatment. At the end of each treatment session, patients were instructed and motivated to perform personal oral hygiene. Moreover, oral hygiene procedures were reinforced at 3 and 6 months after treatment.

After the protocol, patients were enrolled in a maintenance program and recalled for clinical measurements at 1-, 3-, 6-months and 1-year follow-ups. For each patient, a custom-tailored SPT regimen was prescribed to avoid potential mechanical damage at the surgically treated region and enhance plaque reduction using a gentle roll technique for toothbrushing and interproximal cleaning devices.

ELIGIBILITY:
Inclusion Criteria:

* good condition of general health
* a minimum of 2 teeth for each quadrant with
* Pocket Depth (PD) ranging from 4-6 mm
* no involvement of the furcation
* a minimum of six teeth per quadrant, respectively

Exclusion Criteria:

* periodontal therapy during the last 12 months
* assumption of antibiotics during the last 6 months
* pregnancy
* any systemic condition which might affect the effects of the study treatment
* previous or current radiation or immunosuppressive therapies
* use of mouthwash containing antimicrobials during the previous 3 months
* no use of hormonal contraceptives
* medication by anti-inflammatory and immunosuppressive drugs
* previous history of hard drinking
* smoking
* class II and III tooth mobility

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Reduction of Serum C-reactive protein changes | 1-year follow up
  evaluation of serum c-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: Pubmed